CLINICAL TRIAL: NCT04669470
Title: Influence of Bariatric Endoscopy on Clinical Course of NAFLD
Brief Title: Bariatric Endoscopy and NAFLD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Ostrava (Other)
Collaborators: University Hospital Olomouc (Other); University Hospital Ostrava (Other); Palacky University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 08_RVO-FNOs_2020
Record Dates: First submitted 2020-12-09; First posted 2020-12-16 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-11

CONDITIONS: Obesity; NAFLD; Liver Steatosis; Liver Fibrosis
Keywords: Obesity; NAFLD; liver steatosis; liver fibrosis; bariatric endoscopy; weight lose
MeSH Terms: conditions — Obesity; Non-alcoholic Fatty Liver Disease; Fatty Liver; Liver Cirrhosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group with adjustable IGB (Active Comparator)
  Interventions: Procedure: bariatric endoscopy, mainly intragastric baloons, plication of stomach too
- Group with nin-adjustable IGB (Active Comparator)
  Interventions: Procedure: bariatric endoscopy, mainly intragastric baloons, plication of stomach too

INTERVENTIONS:
Procedure: bariatric endoscopy, mainly intragastric baloons, plication of stomach too — bariatric endoscopy, mainly intragastric baloons, plication of stomach too

SUMMARY:
Find out how bariatric endocopy will influence clinical course of non alcoholic fatty liver disease.

DETAILED DESCRIPTION:
The study will test and investigate the impact of bariatric endoscopy (various types of intragastric balloons, endoscopic sleeve gastroplasty, aspiration therapy) on components of the metabolic syndrome in obese patients, especially on influencing non-alcoholic steatosis and steatohepatitis and signs of liver fibrotization and weight reduction. The method consists in performing a mini-invasive endoscopic procedure and, as a result, in reduced food intake.

Current state of knowledge:

Based on data evaluated according to EBM (Evidence Based Medicine), it is an indisputable fact that bariatric methods have a demonstrable effect not only on improving the parameters and regression of many metabolic syndromes, but also improve the course of non-alcoholic fatty liver disease (NAFLD). It is this nosological unit that is becoming the dominant cause of liver disease in developed countries and has two subunits, where simple hepatic steatosis (NAFL) is considered a benign disease, while the second, where fat accumulation in the liver is associated with the inflammatory process called non-alcoholic steatohepatitis (NASH). ) has serious consequences for the liver with the development of fibrotization leading to cirrhosis with all its adverse effects. Recently, however, it has been shown that even simple steatosis is not as benign as it seemed, but carries an independent risk for the patient due to an increased incidence of cardiovascular diseases, oncological manifestations and a higher incidence of metabolic syndrome manifestations. Classical bariatric endoscopy carries a number of risks associated with the patient for the surgical procedure, however, we also have less invasive methods of gradually more and more developing endoscopy and dreams of associated bariatric procedures with many times lower risk for the patient.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for participation in this study, subjects must conform to the following inclusion criteria:

1. Age between 21-64 years;
2. BMI >30 Kg/m2
3. Must be able to comply with all study requirements for the duration of the study as outlined in the protocol. This includes complying with the visit schedule as well as study specific procedures such as: clinical assessment , endoscopy, radiography, as well as laboratory investigations.
4. Must be able to understand and be willing to provide written informed consent.

Exclusion Criteria:

* Subjects meeting any of the following exclusionary criteria cannot be enrolled in the study:

  1. Achalasia and any other esophageal motility disorders
  2. Heart diseases: unstable angina, myocardial infarction within the past year, or heart disease classified within the New York Heart Association's Class III or IV functional capacity.
  3. Hypertension: uncontrolled hypertension during last 3 month
  4. Severe renal, hepatic, pulmonary disease or cancer;
  5. GIT stenosis or obstruction
  6. Pregnancy or breastfeeding
  7. Impending gastric surgery 60 days post intervention;
  8. Currently participating in other study
  9. Celiac disease
  10. History of bariatric surgery
  11. Chronic or recent acute pancreatitis
  12. Type 2 diabetes with insuline medication or type 1 diabetes
  13. Hematologic disease or disease with impairment of hemocoagulation
  14. Decompensated psychiatric disease
  15. Autoimmune disease with chronic glucocorticoid or imunosupressive medications
  16. Uncontroled disease of thyroid gland
  17. Excesive abuse of addictive substances such alcohol or other

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Amount of patients with NAFLD with degree of fibrosis of the liver amog patients undergoing bariatric endoscopy and determine influence of bariatric endoscopy on clinical course of NAFLD and liver fibrosis | 24 months
  Amount of patients with NAFLD with degree of fibrosis of the liver amog patients undergoing bariatric endoscopy and determine influence of bariatric endoscopy on clinical course of NAFLD and liver fibrosis

SECONDARY OUTCOMES:
Influence of bariatric endoscopy on improvements of weight, antropometric, improvements in components of metabolic syndrome | 24 months
  Influence of bariatric endoscopy on improvements of weight, antropometric, improvements in components of metabolic syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Adam Vasura, MD, Study Chair — - Department of gastroenterology, hepatology and pancreatology, Internal clinic, University hospital Ostrava; Evzen Machytka, Study Chair — Department of gastroenterology, hepatology and pancreatology, Internal clinic, University hospital Ostrava
Locations (1):
- Department of gastroenterology, hepatology and pancreatology, Ostrava, Czechia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fakhry TK, Mhaskar R, Schwitalla T, Muradova E, Gonzalvo JP, Murr MM. Bariatric surgery improves nonalcoholic fatty liver disease: a contemporary systematic review and meta-analysis. Surg Obes Relat Dis. 2019 Mar;15(3):502-511. doi: 10.1016/j.soard.2018.12.002. Epub 2018 Dec 6. PMID 30683512
- [Background] Machytka E, Klvana P, Kornbluth A, Peikin S, Mathus-Vliegen LE, Gostout C, Lopez-Nava G, Shikora S, Brooks J. Adjustable intragastric balloons: a 12-month pilot trial in endoscopic weight loss management. Obes Surg. 2011 Oct;21(10):1499-507. doi: 10.1007/s11695-011-0424-z. PMID 21553304
- [Background] Leoni S, Tovoli F, Napoli L, Serio I, Ferri S, Bolondi L. Current guidelines for the management of non-alcoholic fatty liver disease: A systematic review with comparative analysis. World J Gastroenterol. 2018 Aug 14;24(30):3361-3373. doi: 10.3748/wjg.v24.i30.3361. PMID 30122876